CLINICAL TRIAL: NCT03069937
Title: A Phase II Study of Docetaxel Before Medical Castration With Degarelix in Patients With Newly Diagnosed Metastatic Prostatic Adenocarcinoma.
Brief Title: Phase II Study of Docetaxel Before Degarelix in Patients With Newly Diagnosed Metastatic Prostate Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102509; Pro00061532 (Other: MUSC)
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Prostatic Adenocarcinoma
MeSH Terms: interventions — Docetaxel; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Docetaxel + Degarelix (Experimental): Docetaxel (TAXOTERE) will be given for up to 6 cycles every 21 days. During the 5th and 6th cycles, degarelix (Firmagon) will be administered on Cycle 5 day 1 and cycle 6 day 8. After cycle 6, degarelix will continue to be given every 28 days for a 5 more doses, for a total of 7 doses.
  Interventions: Drug: Docetaxel; Drug: Degarelix

INTERVENTIONS:
Drug: Docetaxel — The docetaxel dose is a 75mg/m2 intravenous (given through the vein) injection.
  Other Names: taxotere
Drug: Degarelix — Degarelix will be given as a subcutaneous (given under the skin) injection in the abdomen. The first dose will be a 240mg dose; all other doses will be 80 mg.
  Other Names: Firmagon

SUMMARY:
The purpose of this study is to look at patient outcomes when docetaxel is started prior to ADT with degarelix.

DETAILED DESCRIPTION:
This study will look at two drugs, docetaxel and degarelix, which are both FDA approved for the treatment of prostate cancer. Docetaxel is a standard chemotherapy treatment for metastatic prostate cancer. Degarelix is an androgen deprivation therapy (ADT) agent that decreases the amount of testosterone in the body, which helps to fight tumor growth. Usually, docetaxel is given after ADT. This study will look at how your cancer changes when docetaxel is started before ADT. You are being asked to participate in this study because you have metastatic prostate cancer that can be treated with docetaxel and ADT.

ELIGIBILITY:
INCLUSION CRITERIA Patients eligible for study participation must meet all of the following criteria.

1. Histological or cytological diagnosis of adenocarcinoma of the prostate.
2. Metastatic disease identified via radiographic assessment by CT scans of the chest, abdomen, pelvis, and nuclear bone scan. MRI may be used if deemed necessary by the investigator. See Section 8.5 for more details about radiographic assessment requirements.

   More specifically, patients must have at least one of the following at time of study enrollment:
   1. Any visceral metastases identified by CT scans or MRI.
   2. Site(s) of bony metastasis identified by nuclear bone scan, MRI, and/or CT scan.
   3. Lymph node based disease not considered to be within a single radiation therapy port (e.g. at or above the aortic bifurcation.)
3. Non-castrate testosterone level, >50 ng/dl, at study enrollment.
4. Age greater than or equal to 18 years.
5. ECOG performance status 0-2.
6. Meet the following hematologic criteria within 14 days of enrollment to trial:

   1. Absolute neutrophil count > 1,500/mm3
   2. Hemoglobin > 8.0 g/dl (may be transfused)
   3. Platelet count > 100,000 mm3
7. Have adequate end-organ function as defined by the following parameters. All lab values must be obtained within 14 days of enrollment to trial:

   1. Creatinine clearance of > 30 ml/min. Creatinine clearance should be determined by the Cockcroft-Gault formula (Appendix A)
   2. AST < 2 x institutional ULN
   3. ALT < 2 x institutional ULN
   4. Total bilirubin < institutional ULN
8. Agree to use barrier methods of birth control during the docetaxel portion of the protocol and for at least one month after last docetaxel administration.
9. Informed and must sign and give written informed consent in accordance with institutional and federal guidelines.

EXCLUSION CRITERIA

Patients eligible for study participation CANNOT meet any of the following criteria:

1. CNS metastases (brain or leptomeningeal).
2. Osseous metastases felt in the opinion of the clinician to be high-risk for impending pathologic fracture or spinal cord compression.
3. Active cardiac disease defined as symptomatic congestive heart failure, history of NYHA Class III or IV Heart Failure, uncontrollable supraventricular arrhythmias, any history of a ventricular arrhythmia, active angina pectoris, myocardial infarction or coronary intervention within 6 months of registration.
4. Prior malignancy requiring systemic therapy within the last 5 years except for treated basal or squamous cell skin cancer. History of low-grade malignancies with limited potential to progress as determined by the primary investigator may be enrolled.
5. Subjects must not have received any previous androgen deprivation therapy (LHRH agonist or LHRH antagonist) or cytotoxic therapy for prostate cancer in the metastatic setting.

   Exception Patients may have received no more than 30 days of anti-androgen (e.g. bicalutamide) in the metastatic setting prior to the start of study treatment.
6. Subjects must not have had more than 36 months of hormonal therapy in combination with prostatectomy or radiation in the setting of localized disease and must not have shown any evidence of disease recurrence within 12 months after stopping hormonal therapy. Disease recurrence after hormonal therapy is defined as PSA > 0.2ng/dl after prostatectomy + hormonal therapy or PSA that is 2.0ng/dl more than the PSA nadir after radiotherapy + hormonal therapy. Previous hormonal therapy to the prostate must have stopped at least 12 months prior to enrollment.
7. Subjects must not have been treated with prior docetaxel in the setting of metastatic prostate cancer. Subjects may have been treated with docetaxel in the setting of localized prostate cancer (likely as a trial-based neoadjuvant or adjuvant approach to prostatectomy or radiation.) Subjects treated with this approach must not have shown any evidence of disease recurrence within 12 months after stopping docetaxel. Disease recurrence after docetaxel is defined as PSA > 0.2ng/dl after prostatectomy + docetaxel or PSA that is 2.0ng/dl more than the PSA nadir after radiotherapy +docetaxel. Previous docetaxel in the setting of localized prostate cancer must have stopped at least 12 months prior to study enrollment.
8. Palliative radiation therapy may have been received but not within the 30 days prior to study treatment.
9. Presence of peripheral neuropathy > Grade 1.
10. Known HIV-positive
11. Presence of any severe or uncontrolled concurrent medical condition felt in the opinion of the investigator to increase the risk of serious toxicity from the study therapy.
12. Prior hypersensitivity to any of the components of the study drugs.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2024-12-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 52 subjects in the study, 51 were evaluable for the primary endpoint. The one unevaluable subject got a second primary malignancy noted after registration but prior to start of study.
Period: Overall Study
Arm/Group | Docetaxel + Degarelix
Started | 52
Completed | 51
Not Completed | 1
Not completed — Second primary malignancy noted | 1

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel + Degarelix
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (7.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: PSA Response at 10 Months
Description: PSA complete response is defined as PSA level less than or equal to 0.2 ng/ml for two consecutive measurements at least three weeks apart. Date of complete response will be defined as the date of first recorded value less than 0.2 ng/ml. PSA progression will be defined as > 25% increase from the PSA nadir (lowest PSA value recorded since trial enrollment) and > 2 ng/dl above the nadir. Two consecutive increases must be recorded at least three weeks apart. Date of PSA progression will be defined as the first recorded PSA value that is a > 25% increase from the PSA nadir and > 2 ng/dl above the nadir.
Time Frame: 10 months
Population: The Primary endpoint for this trial is a binary indicator of PSA less than or equal to 0.2 ng/mL at 10 months (40 weeks) on study. This also represents 7 months (28 weeks) on androgen deprivation therapy with Degarelix
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel + Degarelix
Number analyzed (Participants) | 51
Participants | 15

2. Secondary Outcome: PSA Response at 6 Months
Description: as for outcome 1
Time Frame: 6 months
Population: Undetectable PSA at 6 months is a binary indicator for each patient of PSA less than or equal to 0.2 ng/dl at 6 months (24 weeks) on study.
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel + Degarelix
Number analyzed (Participants) | 51
Participants | 14

3. Secondary Outcome: Number of Grade 3 and 4 Adverse Events Related to Docetaxel During First 4 Cycles
Description: This measure reports the number of Grade 3 and 4 adverse events that were possibly or probably related to docetaxel and occurred during the first 4 cycles (approximately 12 weeks) of treatment
Time Frame: Up to 12 weeks (first 4 cycles of docetaxel)
Population: Total possibly and probably related events that occur in the first 4 cycles Docetaxel
Measure: Count of Units; unit: adverse events
Units Other Than Participants: adverse events
Arm/Group | Docetaxel + Degarelix
Number analyzed (Participants) | 51
Number analyzed (adverse events) | 273
adverse events | 6

4. Secondary Outcome: Frequency of Disease Progression at 12 Weeks Using PSA
Description: PSA progression will be defined as > 25% increase from the PSA nadir (lowest PSA value recorded since trial enrollment) and > 2 ng/dl above the nadir. Two consecutive increases must be recorded at least two weeks apart. Date of PSA progression will be defined as the first recorded PSA value that is a > 25% increase from the PSA nadir and > 2 ng/dl above the nadir. PSA progression will not be established during the first 12 weeks of therapy (4 cycles of docetaxel) as defined by PCWG2 criteria. Thus subjects with no PSA decline from baseline during therapy will have date of PSA progression defined as first PSA value after 12 weeks that is a > 25% increase from the PSA nadir and > 2 ng/dl above the nadir.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel + Degarelix
Number analyzed (Participants) | 51
Participants | 12

5. Secondary Outcome: PSA Response at 12 Weeks
Description: PSA complete response is defined as PSA level less than or equal to 0.2 ng/ml for two consecutive measurements at least two weeks apart. Date of complete response will be defined as the date of first recorded value less than 0.2 ng/ml.
  PSA Partial Response is defined as a decline of PSA from trial baseline of > 50% for two consecutive measurements at least two weeks apart. Date of partial response will be defined as the date of first recorded decline of > 50% baseline.
  PSA progression is defined in outcome 4.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel + Degarelix
Number analyzed (Participants) | 51
Participants
  PSA complete response | 1
  PSA partial response | 20

6. Secondary Outcome: Time to Development of Castration Resistance After Initiation With ADT
Description: This will be defined as the time from initial Degarelix injection to the time of disease progression (clinical, radiographic or PSA. Determination of castration resistant disease status will require disease progression and a measured serum testosterone level less than 50 ng/dl.
Time Frame: From initiation of Degarelix until disease progression or end of follow-up (up to 34 months)
Population: evaluable subjects who were administered Degarelix
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel + Degarelix
Number analyzed (Participants) | 40
months | 16.1 [9.73 to 23.5]

7. Secondary Outcome: Progression Free Survival
Description: Progression free Survival (PFS) will be defined as the duration of time from start of study treatment to time of disease progression or death, whichever comes first.
Time Frame: 34 months
Population: progressions from day 1 of Docetaxel
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel + Degarelix
Number analyzed (Participants) | 41
months | 15.9 [11.4 to 24.2]

8. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time interval from trial enrollment to death due to any cause. Survival times will be censored for patients lost to follow-up or still alive at the trial's termination.
Time Frame: From trial enrollment until death or end of follow-up (up to 52.4 months)
Population: subjects who died from any cause
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel + Degarelix
Number analyzed (Participants) | 28
months | 52.4 [46.9 to 57.9]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed up to 10 months. All-cause mortality was assessed up to 52.4 months.
Arm/Group | Docetaxel + Degarelix
All-Cause Mortality (participants affected / at risk) | 28/51
Serious Adverse Events (participants affected / at risk) | 4/51
Other Adverse Events (participants affected / at risk) | 49/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel + Degarelix (N=51)
febrile neutropenia (Blood and lymphatic system disorders) | 1
myositis (Musculoskeletal and connective tissue disorders) | 1
Anorectal infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1 — pneumonia
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel + Degarelix (N=51)
Fatigue (General disorders) | 39
Hot flashes (Vascular disorders) | 29
Alopecia (Skin and subcutaneous tissue disorders) | 26
Nausea (Gastrointestinal disorders) | 18
Edema limbs (General disorders) | 17
Constipation (Gastrointestinal disorders) | 16
Dysgeusia (Nervous system disorders) | 16
Nail discoloration (Skin and subcutaneous tissue disorders) | 16
Injection site reaction (General disorders) | 14
Watering eyes (Eye disorders) | 11
Diarrhea (Gastrointestinal disorders) | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Hypertension (Vascular disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 6
Pain (General disorders) | 5
Weight loss (Investigations) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Rash maculo papular (Skin and subcutaneous tissue disorders) | 5
Flu like symptoms (General disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 4
Insomnia (Psychiatric disorders) | 4
Hypotension (Vascular disorders) | 4
Peripheral motor neuropathy (Nervous system disorders) | 3
Cystitis noninfective (Renal and urinary disorders) | 3
Nail infection (Infections and infestations) | 3
Abdominal pain (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 3
Paresthesia (Nervous system disorders) | 3
Hematuria (Renal and urinary disorders) | 3
Urinary retention (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT03069937/Prot_SAP_001.pdf